CLINICAL TRIAL: NCT00384670
Title: A Phase I/II Trial of a Tetravalent Live Attenuated Dengue Vaccine in Flavivirus Antibody Naïve Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WRAIR 1048; HSRRB#A-12189 (Other: USAMRMC); GSK Dengue-003 (Other: GSK)
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-01

CONDITIONS: Dengue Fever
Keywords: dengue; vaccine
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dengue and Japanese Encephalitis vaccine (Experimental): 1 mL subcutaneous injection Dengue Vaccine Formulation 17 on Day 0 and Day 60. 0.5 mL subcutaneous injection Licensed Japanese Encephalitis (JE) Vaccine on months 7 and 7.5.
  Interventions: Biological: Dengue Vaccine Formulation 17; Biological: Licensed Japanese Encephalitis (JE) Vaccine

INTERVENTIONS:
Biological: Dengue Vaccine Formulation 17 — Tetravalent live attenuated DEN vaccine candidate. Containing dengue serotypes 1,2, and 3 vaccines produced at the Salk Institute and dengue serotype 4 produced at the WRAIR Pilot Bioproduction Facility. Dosage 1 mL administered via injection at Day 0 and Day 60.
  Other Names: F17
Biological: Licensed Japanese Encephalitis (JE) Vaccine — Produced by the Thailand GPO using a Beijing strain of JE in liquid form; dosed at 0.5 mL ot 7 and 7.5 months.
  Other Names: JE

SUMMARY:
To assess the safety, reactogenicity and immunogenicity of two doses of the dengue vaccine in Flavi-virus antibody-naive children between 6 and 9 years of age.

DETAILED DESCRIPTION:
This study was a Phase I/II, open-label trial with one treatment group; 7, healthy, flavivirus naïve children between the ages of 6 and 7 years residing in Bangkok, Thailand. Seronegative status was determined by measuring neutralizing (N) antibody titers to dengue 1-4 and JE virus (JE) using hemagglutination inhibition (HAI) (1st) and PRNT (2nd) assays. Titers <10 and <10, respectively, were considered negative. Enrolled children received two doses of tetravalent dengue vaccine at study months 0 and 6, and two doses of JE vaccine (study benefit) at study months 7 and 7.5. Enrolled children attended 20 study visits, received 4 injections, and 7 venipunctures (one additional blood sample for screening). In the acute period (1 month) following vaccination, safety was assessed using symptom diary cards and clinical and laboratory evaluations. Viremia was measured 10 days post dengue vaccination. Solicited and unsolicited adverse events were assessed for 30 days following each dengue vaccination. Serious adverse events were assessed throughout the study period. In the case of illness, investigators would complete additional clinical and virologic evaluations. Dengue vaccine immunogenicity was assessed 30 days following each dengue vaccination using the PRNT50 assay. The According to Protocol (ATP) cohort was determined by evaluating the occurrence of intermittent natural dengue infection using ELISA IgM/IgG titer ratios. A long-term follow-up of dengue vaccine recipients is described in a separate protocol (Dengue-005 protocol).

ELIGIBILITY:
Inclusion Criteria:

* A male or female child six to nine years of age (greater than or equal to 6 years of age and less than 10 years of age) at the time of the first vaccination.
* Free of obvious health problems as established by medical history and physical examination before entering into the study.
* Seronegative by HAI and screening PRNT for antibodies to dengue types 1-4 and Japanese Encephalitis (JE) virus
* Written informed consents by the parent of the subject for screening and enrollment into the study.

Exclusion Criteria:

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned administration during the study (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Use of any investigational or non-registered drug or vaccine other than the protocol-specified vaccines within 30 days preceding the administration of the first dengue vaccine dose or planned use during the study period.
* Planned administration of a vaccine not foreseen by the study protocol and within 30 days prior or after any dengue/JE vaccine administration.
* Any current medical condition determined to be serious by the investigator (e.g. seizures)
* History of chronic headaches or a first order family member (parent or sibling) with a history of chronic headaches
* Abnormal clinical laboratory screening test result (based on normal values set by the laboratory) that is deemed clinically significant by the investigator or Medical Monitor (including seropositivity for HBsAg or anti-HCV)
* Previous vaccination against yellow fever virus, JEV, or tick-borne encephalitis virus (TBE) or existence of any flavivirus antibody
* Any suspected or confirmed immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Family history of a congenital or hereditary immunodeficiency
* Acute illness at time of enrollment (defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhea or mild upper respiratory infection without fever, i.e., oral temperature <37.5°C.
* Administration of immunoglobulins and/or blood products within 6 months prior to study entry or planned administration during the study period
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines (including neomycin, streptomycin, gentamicin, amikacin, tobramycin, kanamycin and bacitracin; allergy to dogs or monkeys or hypersensitivity to proteins of rodent or neural origin or to thimerosal, allergy to porcine gelatin)
* Child whose parent has no easy access to a fixed or mobile telephone
* Plans to move from Bangkok during the first 8.5 months after initial vaccination
* Parental illiteracy.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2003-08; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MAJ Stephen J Thomas, MD, Principal Investigator — Department of Virology USAMC-AFRIMS; Sriluck Simasathien, MD, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Department of Pediatrics, Pharamongkutklao Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Simasathien S, Thomas SJ, Watanaveeradej V, Nisalak A, Barberousse C, Innis BL, Sun W, Putnak JR, Eckels KH, Hutagalung Y, Gibbons RV, Zhang C, De La Barrera R, Jarman RG, Chawachalasai W, Mammen MP Jr. Safety and immunogenicity of a tetravalent live-attenuated dengue vaccine in flavivirus naive children. Am J Trop Med Hyg. 2008 Mar;78(3):426-33. PMID 18337339

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dengue Vaccine and Japanese Encephalitis Vaccine: 1 mL subcutaneous injection Dengue Vaccine Formulation 17 on Day 0 and Day 60. 0.5 mL subcutaneous injection Licensed Japanese Encephalitis (JE) Vaccine on months 7 and 7.5.
Arm/Group | Dengue Vaccine and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.6 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  Thailand | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Solicited Adverse Events Within 21 Days After the First Dose of Dengue Vaccine.
Description: Number of solicited general symptoms within the 21-day follow-up after dengue dose 1 (total vaccinated cohort).
Time Frame: 21 days
Measure: Number; unit: adverse events
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
adverse events
  Abdominal Pain | 1 [0.4 to 57.9]
  Fatigue | 3 [9.9 to 81.6]
  Headache | 5 [29.0 to 96.3]
  Muscle and/or Joint Aches | 3 [9.9 to 81.6]
  Pain Behind Eyes | 2 [28.6 to 3.7]
  Photophobia | 0 [0 to 41.0]
  Pruritus | 2 [3.7 to 71.0]
  Elevated Temperature | 4 [18.4 to 90.1]
  Vomiting and/or Nausea | 1 [0.4 to 57.9]

2. Secondary Outcome: Number of Unsolicited Adverse Events Within 30 Days After Each Dose of Dengue Vaccine
Description: Number of subjects with unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term, within 30 days after dengue vaccine (total vaccinated cohort)
Time Frame: 30 days
Measure: Number; unit: adverse events
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
adverse events
  At least one symptom | 7 [59.0 to 100]
  Infections and Infestations | 2
  Nervous System Disorders | 1
  Respiratory, Thoracic and Mediastinal Disorders | 6

3. Secondary Outcome: Number of Solicited Adverse Events for 21 Days (0-20) After the Second Dose of Dengue Vaccine
Description: Number of solicited general symptoms within the 21-day follow-up of dengue dose 2 vaccine dose (total vaccinated cohort)
Time Frame: 21 Days (0-20) After the Second Dose of Dengue Vaccine
Measure: Number; unit: adverse events
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
adverse events
  Abdominal Pain | 0
  Fatigue | 3
  Headache | 3
  Muscle and/or Joint Aches | 2
  Pain Behind Eyes | 1
  Photophobia | 1
  Pruritus | 2
  Elevated Temperature | 3
  Vomiting and/or Nausea | 1

4. Secondary Outcome: Percentage of Individuals With Neutralizing Antibody (Seroconversion) to Japanese Encephalitis (JE) and 4 Dengue Types, 30 Days After the Second Dose of JE Vaccine.
Description: Percentage of individuals with ≥ 10 dilution (DIL) for neutralizing (N) Ig to DEN-1, N Ig to DEN-2, N Ig to DEN-3, N Ig to DEN-4, and N Ig to Japanese encephalitis (JE) vaccine antibody titers.
Time Frame: 30 days after the second dose of JE vaccine
Population: 1 subjects experience an asymptomatic, sub-clinical, DEN-2 virus infection prior to dengue vaccine dose 1 and was eliminated from the according to protocol (ATP) analysis of immunogenicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 6
percentage of participants
  N Ig to DEN-1 | 100 [54.1 to 100]
  N Ig to DEN-2 | 100 [54.1 to 100]
  N Ig to DEN-3 | 100 [54.1 to 100]
  N Ig to DEN-4 | 83.3 [35.9 to 99.6]
  N Ig to JE | 33.3 [4.3 to 77.7]

5. Secondary Outcome: Neutralizing Antibody (GMT) to JE and 4 Dengue Types, 30 Days After the Second Dose of JE Vaccine.
Description: Geometric mean titers (GMT) for neutralizing (N) Ig to DEN-1, N Ig to DEN-2, N Ig to DEN-3, N Ig to DEN-4, and N Ig to JE vaccine antibody titers.
Time Frame: Approximately Day 225 and Day 255
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 6
titer
  N Ig to DEN-1 | 55.8 [15.3 to 203.1]
  N Ig to DEN-2 | 107.4 [39.5 to 292.0]
  N Ig to DEN-3 | 37.0 [8.7 to 158.2]
  N Ig to DEN-4 | 36.9 [11.0 to 123.4]
  N Ig to JE | 8.7 [3.4 to 22.5]

6. Secondary Outcome: Number of Solicited Symptoms 7 Days (0-6) After First Dose of Japanese Encephalitis (JE) Vaccine.
Description: Number of solicited general symptoms within the 7-day follow-up after the first dose of Japanese encephalitis (JE) vaccine doses (total vaccinated cohort)
Time Frame: Approximately Day 225 and Day 255
Measure: Number; unit: adverse events
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
adverse events
  Abdominal Pain | 1
  Fatigue | 1
  Headache | 2
  Muscle and/or Joint Aches | 1
  Photophobia | 1
  Pruritus | 1
  Elevated Temperature | 1
  Vomiting and/or Nausea | 1

7. Secondary Outcome: Number of Solicited Symptoms 7 Days (0-6) After Second Dose of Japanese Encephalitis (JE) Vaccine.
Description: Number of solicited general symptoms within the 7-day follow-up after the second dose of Japanese encephalitis (JE) vaccine doses (total vaccinated cohort)
Time Frame: Approximately Day 225 and Day 255
Measure: Number; unit: Number of solicited general symptoms
Arm/Group | Dengue and Japanese Encephalitis Vaccine
Number analyzed (Participants) | 7
Number of solicited general symptoms
  Abdominal Pain | 0
  Fatigue | 0
  Headache | 1
  Muscle and/or Joint Aches | 0
  Photophobia | 0
  Pruritus | 1
  Elevated Temperature | 0
  Vomiting and/or Nausea | 0

ADVERSE EVENTS:
Arm/Group | Dengue Vaccine and Japanese Encephalitis Vaccine
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 0.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dengue Vaccine and Japanese Encephalitis Vaccine (N=7)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Headache (Nervous system disorders) | 5 (8)
Muscle and/or joint aches (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain behind eyes (Eye disorders) | 3 (3)
Photophobia (Eye disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Elevated Temperature (General disorders) | 5 (7)
Vomiting and/or Nausea (Gastrointestinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Meibomian cyst infected (Infections and infestations) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No